CLINICAL TRIAL: NCT03732365
Title: A Phase 2 Randomized Study to Compare the Efficacy and Safety of Ultrasonic Drug Delivery to Standard of Care for the Treatment of Acute Bacterial Skin and Skin Structure Infections in Chronic Non-Healing Wounds
Brief Title: Phase 2 Randomized Study to Compare Ultrasonic Drug Delivery to Standard of Care for the Treatment of Infections in Non-Healing Wounds
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sonescence, Inc. (Industry)
Collaborators: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SON2018-001
Record Dates: First submitted 2018-10-25; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Acute Bacterial Skin and Skin Structure Infection (ABSSSI); Non-healing Wound
MeSH Terms: interventions — Cefazolin

STUDY DESIGN:
Intervention Model Description: Single-center, parallel-group study to compare the efficacy and safety of UDD plus standard of care with standard of care alone for the treatment of skin and soft tissue infections in chronic non-healing wounds.
Who Masked: Outcomes Assessor
Masking Description: This study will be observer-blinded. Each investigational site will be required to have a Sponsor-approved plan (a site-specific Blinding Plan) that describes site-specific precautions being taken to ensure that the study is observer-blinded, taking into account the specific subject care procedures, equipment, and information accessibility at that site. At each investigational site, at least 1 blinded investigator (referred to as "Blinded Observer") will not know the subject's treatment assignment and will conduct clinical assessments (including efficacy and safety. The Blinded Observer will not ask other members of the study team, the subject, or the subject's parent(s)/legally acceptable representative(s) which study treatment is being given, and will avoid all attempts to uncover treatment assignment. The Blinded Observer will see the subject during times when study treatment is NOT being administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Investigational Group (Experimental): Patients who are randomized to the investigational regimen will receive Ultrasonic Drug Delivery, which includes infusion of up to 2 grams of cefazolin in 100 mL saline followed by external ultrasound in addition to standard of care antibiotic treatment according to the antibiotic package insert instructions for the particular gram-positive pathogen over a period of no more than 14 days as well as standard of care adjunct therapy.
  Interventions: Combination Product: Ultrasonic Drug Delivery
- Comparator Group (Active Comparator): Patients who are randomized to the comparator regimen will receive antibiotic according to the antibiotic package insert instructions for standard of care for the particular gram-positive pathogen over a period of no more than 14 days as well as standard of care adjunct therapy.
  Interventions: Drug: Standard of Care Antibiotic Treatment

INTERVENTIONS:
Combination Product: Ultrasonic Drug Delivery — A maximum dose of 2 grams cefazolin in a solution of 1 gram/100 mL sterile saline will be injected into the affected area, followed by a 3-minute application of external ultrasound delivered at an acoustic intensity equal to 3 watts/square centimeter of surface area.
  Other Names: Cefazolin with external ultrasound
  Arms: Investigational Group
Drug: Standard of Care Antibiotic Treatment — Antibiotic treatment according to the antibiotic package insert instructions for the particular gram-positive pathogen over a period of no more than 14 days.
  Arms: Comparator Group

SUMMARY:
This is a randomized study to compare the safety and efficacy of a single dose of up to 2 grams of cefazolin administered using a new drug delivery method called Ultrasonic Drug Delivery (UDD), combined with standard of care (SOC) antibiotic therapy, oral or IV, compared to standard of care (SOC) antibiotic therapy alone, in treating chronic wounds with skin and soft tissue infection, containing gram-positive pathogens, in lower extremities.

DETAILED DESCRIPTION:
This is a Phase 2, single-center, parallel-group study to compare the efficacy and safety of UDD plus standard of care (SOC) with SOC alone for the treatment of skin and soft tissue infections in non-healing wounds. After review of screening results to determine eligibility, a patient will be randomly assigned to one of the two treatments:

Investigational Group: This group will receive administration of a single dose of cefazolin, using a novel new drug delivery system called Ultrasonic Drug Delivery (UDD), to the site of infection, combined with SOC, followed by best available adjunct therapy. An optional two additional treatments will be available if needed.

Comparator Group: This group will receive conventional standard of care treatment followed by best available adjunct therapy.

Efficacy will be assessed by clinical response based on the presence of vascularized granulation tissue, reduction of pain, temperature, measurement of lesion size and temperature, culture and gram stain results, and clinical signs of infection (erythema, induration/swelling, fluctuance, purulent drainage, warmth/localized heat, and tenderness/pain). Additionally, efficacy will be assessed by resolution of infection and microbiological assessments.

Safety will be assessed by reported adverse events, clinical laboratory tests (hematology, serum chemistry, fasting glucose, hs-CRP), and concomitant medication.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Must have a non-healing wound which shows clinical signs of infection characterized by erythema and at least two of the following signs of infection: Induration/swelling; Purulent drainage/discharge; Fluctuance; Heat/localized warmth; Tenderness/pain to palpation
* Patient must have one (1) or more of the following confirmed infection types of the lower extremity: a) Cellulitis/erysipelas: A diffuse skin infection characterized by spreading areas of redness, edema, and/or induration; b) Wound infection: An infection characterized by purulent drainage from a wound with surrounding redness, edema, and/or induration; c) Major cutaneous abscess: An infection characterized by a collection of pus within the dermis or deeper that is accompanied by redness, edema, and/or induration
* A minimum affected area that involves: At least 75cm2 of erythema; and is defined by a margin of erythema in at least one (1) direction that is ≥ 5 cm from the edge of the wound.
* In addition to the requirement for erythema, all patients are required to have at least two (2) of the following signs of acute bacterial skin and skin structure infection (ABSSSI): a) Purulent drainage/discharge; b) Fluctuance; c) Heat/localized warmth; d) Tenderness to palpation; and e) Swelling/induration
* Patients must present with at least ONE (1) of the following systemic signs of infection: a) An elevated body temperature ≥ 100.4 Fahrenheit as measured by clinical staff or investigator within 24 hours of baseline at screening; and/or b) White blood cell count > 12,000 cells/mm3; c) manually performed white blood differential count with ≥ 10% band forms, regardless of peripheral white blood cell count.
* Bacteria culture positive for gram positive bacteria.
* Ability and willingness to accept subcutaneous administration of antibiotic and local anesthesia.
* For females of reproductive potential: use of highly effective contraception and agreement to use such a method during study participation.
* Agreement to adhere to the study intervention regimen.

Exclusion Criteria:

* Patients with conditions that would alter the interpretation of a primary endpoint, including: patients with neutropenia; and/or patients with peripheral neuropathy
* Participation in another study of an investigational drug or device within 30 days prior to administration of investigational treatment.
* Pregnant or lactating women.
* Patients with a known allergic reaction or hypersensitivity to cefazolin or penicillin.
* Infections caused exclusively by gram-negative bacteria (without gram-positive bacteria present) and infections caused by fungi, whether alone or in combination with a bacterial pathogen.
* Presence of gram-negative bacteremia, even in the presence of gram-positive infection or gram-positive bacteremia.
* Patients with evidence of meningitis, gas gangrene, gangrene, septic arthritis, or osteomyelitis, endovascular infection, such as clinical and/or echocardiographic evidence of endocarditis or septic thrombophlebitis.
* Infections involving a diabetic foot ulceration, perirectal abscess or a decubitus ulcer.
* Patients with an infection involving a limb with evidence of critical ischemia of an affected limb defined as any of the following criteria: absent or abnormal Doppler wave forms, toe blood pressure of <45 mm Hg, ankle brachial index <0.4, critical ischemia as assessed by a vascular surgeon.
* Patient with an infected device.
* Suspicion of skin cancer at the wound site (i.e., clinical evaluation is currently on-going).
* Patients who have a history of clinically significant or uncontrolled cardiac disease, including congestive heart failure, angina, myocardial infarction, arrhythmia, including New York Heart Association (NYHA) functional classification of III (marked limitation of physical activity comfortable at rest but less than ordinary activity results in fatigue, palpitation or dyspnoea) or Class IV (unable to carry out any physical activity without discomfort - symptoms at rest. If any physical activity is undertaken, discomfort is increased).
* Patients who have any other life-threatening illness or organ system dysfunction, which, in the opinion of the Investigator, would either compromise patient safety or interfere with the evaluation of the safety of the test drug.
* Anticipated need of antibiotic therapy for longer than 14 days.
* Medical conditions in which chronic inflammation may preclude assessment of clinical response to therapy even after successful treatment (e.g., chronic stasis dermatitis of the lower extremity).
* Known or suspected human immunodeficiency virus (HIV) infected patients with a CD4 (cluster of differentiation 4) cell count < 200 cells/mm3 or with a past or current acquired immunodeficiency syndrome (AIDS) - defining condition and unknown CD4 count.
* Patients with a recent bone marrow transplant.
* Patients receiving oral steroids > 20 mg prednisone per day (or equivalent) or receiving immunosuppressant drugs after organ transplantation.
* Patients with a rapidly fatal illness who are not expected to survive for three months.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Wound healing and eligibility for grafting | 12 weeks
  Number of wounds 100% granulation/ready to graft as assessed by a blinded observer
Reduction or elimination of pain | 12 weeks
  Pain assessed by participant questionnaire

SECONDARY OUTCOMES:
Clinical signs and symptoms of infection will be assessed | Day 9 and Day 91
  Eradication of infection; percent of wound closure

CONTACTS AND LOCATIONS:
Overall Officials: David G Armstrong, Ph.D., DPM, Principal Investigator — University of Southern California